CLINICAL TRIAL: NCT03291821
Title: Double Ovarian Stimulation in Cases of Preimplantation Genetic Testing: Comparison of Embryo Quantity and Embryonic Quality Using MitoScore
Brief Title: DuoStim in Cases of PGT: Comparison of Embryo Quantity and Embryonic Quality Using MitoScore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1702-MAD-014-MC
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Infertility, Female
Keywords: DuoStim; MitoScore; Preimplantation genetic diagnosis; MII oocyte
MeSH Terms: conditions — Infertility, Female | interventions — Menotropins; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; ganirelix; cetrorelix; Gonadotropin-Releasing Hormone; Triptorelin Pamoate; Sperm Injections, Intracytoplasmic; Embryo Transfer; Pregnancy Tests

STUDY DESIGN:
Intervention Model Description: Unicentric, prospective, randomized, non-blind, parallel-group controlled phase IV clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DuoStim (Experimental): Two controlled ovarian stimulation within the same menstrual cycle using human menopausal gonadotropin 225 IU/day subcutaneously, GnRH antagonist in a dose of 0.25 mg/day subcutaneously and 0.2 mg of GnRH analog to induce oocyte maturation. It will be followed by ovarian puncture, oocyte isolation, intracytoplasmic sperm injection and trophectoderm biopsy at the blastocyst stage. Preimplantation genetic test and MitoScore will be performed in all the embryos prior to the embryo transfer. At this step embryos will be frozen to wait for the results. Chromossomally normal embryos will be thawed and transferred to the uterus in a deferred cycle. A pregnancy test will be performed when appropriate.
  Interventions: Drug: human menopausal gonadotropin; Drug: GnRH antagonist; Drug: GnRH analog; Procedure: Trophectoderm biopsy; Diagnostic Test: MitoScore; Procedure: Intracytoplasmic sperm injection; Procedure: Ovarian puncture; Diagnostic Test: Preimplantation genetic test; Procedure: Embryo transfer; Diagnostic Test: Pregnancy test; Procedure: Embryo freezing; Procedure: Embryo thawing
- Conventional Stimulation (Active Comparator): Two controlled ovarian stimulation in different menstrual cycles using human menopausal gonadotropin 225 IU/day subcutaneously, GnRH antagonist in a dose of 0.25 mg/day subcutaneously and 0.2 mg of GnRH analog to induce oocyte maturation. It will be followed by ovarian puncture, oocyte isolation, intracytoplasmic sperm injection and trophectoderm biopsy at the blastocyst stage. Preimplantation genetic test and MitoScore will be performed in all the embryos prior to the embryo transfer. At this step embryos will be frozen to wait for the results. Chromossomally normal embryos will be thawed and transferred to the uterus in a deferred cycle. A pregnancy test will be performed when appropriate.
  Interventions: Drug: human menopausal gonadotropin; Drug: GnRH antagonist; Drug: GnRH analog; Procedure: Trophectoderm biopsy; Diagnostic Test: MitoScore; Procedure: Intracytoplasmic sperm injection; Procedure: Ovarian puncture; Diagnostic Test: Preimplantation genetic test; Procedure: Embryo transfer; Diagnostic Test: Pregnancy test; Procedure: Embryo freezing; Procedure: Embryo thawing

INTERVENTIONS:
Drug: human menopausal gonadotropin — human menopausal gonadotropin subcutaneously
  Other Names: menopur; meriofert
Drug: GnRH antagonist — GnRH antagonist subcutaneously
  Other Names: orgalutran; cetrotide
Drug: GnRH analog — GnRH analog subcutaneously
  Other Names: decapeptyl
Procedure: Trophectoderm biopsy — Trophectoderm biopsy is the process of removing few cells from an in vitro fertilization embryo.
  Other Names: embryo biopsy; blastocyst biopsy
Diagnostic Test: MitoScore — The cells removed from an in vitro fertilization embryo during the trophectoderm biopsy will be used to assess the mitochondrial DNA content as a viability indicator in the euploid embryos.
Procedure: Intracytoplasmic sperm injection — ICSI is an in vitro fertilization procedure in which a single sperm is injected directly into an oocyte.
  Other Names: ICSI
Procedure: Ovarian puncture — Egg retrieval is a simple procedure. It is performed in an operating room for safety reasons. It is performed vaginally and involves aspirating the follicular fluid through a thin needle. Embryologists then retrieve from this fluid the eggs that have matured during stimulation. It lasts for 5 to 15 minutes, and a mild sedative is administered to prevent any kind of pain during the procedure.
  Other Names: pick up; egg retrieval
Diagnostic Test: Preimplantation genetic test — The cells removed from an in vitro fertilization embryo during the trophectoderm biopsy will be tested for chromosomal normalcy before transferring the embryo to the uterus.
Procedure: Embryo transfer — Embryo transfer refers to a step in the process of assisted reproduction in which embryos are placed into the uterus
Diagnostic Test: Pregnancy test — A pregnancy test is used to determine whether a woman is pregnant.
Procedure: Embryo freezing — Embryo freezing is a method for cryopreserving embryos.
  Other Names: embryo cryopreservation; embryo vitrification
Procedure: Embryo thawing — Embryo thawing is the procedure to recover previously frozen embryos prior to an embryo transfer.

SUMMARY:
Since preimplantation genetic testing (PGT) is being more frequently requested from patients as women pursue infertility treatments at an advanced age with a poorer prognosis, sometimes physicians are compelled to perform several stimulation cycles to obtain more eggs and, consequently, a greater number of biopsied embryos. Hence, the idea of carrying out this study arises as an attempt to optimize each menstrual cycle to the maximum.

It is believed that the double stimulation (DuoStim) protocol could be an alternative for this group of patients, allowing to obtain a larger number of oocytes in a shorter period, thus, increasing the number of biopsied embryos and possibly decreasing the interval to achieve a successful pregnancy.

The investigators aim to evaluate the potential usefulness of the DuoStim protocol for patients desiring to obtain oocytes as soon as possible. Using PGT, the investigators will compare the rate of euploid embryos per cycle in patients undergoing DuoStim protocol versus patients undergoing two conventional controlled ovarian hyperstimulation in consecutive cycles. Patients will include women with advanced age and poor response.

This is a unicentric, prospective, randomized, non-blind, parallel-group controlled phase IV clinical study. The investigators hypothesize that the rate of euploid embryos per cycle is similar in the DuoStim group compared to the group undergoing two conventional controlled ovarian hyperstimulation in consecutive cycles.

Furthermore the investigators will evaluate if there are differences regarding the number of total oocytes obtained, the number of mature oocytes, the number of biopsied blastocysts and the MitoScore index of the available euploid embryos.

DETAILED DESCRIPTION:
Classically, the follicular development was thought to occur only during the follicular phase of the menstrual cycle. However, new data demonstrated several waves of cyclic development of the antral follicles within the same menstrual cycle. Some authors insist that follicles formed during the luteal phase may have a similar ovulation potential of those formed in the follicular phase, thus offering new possibilities for ovarian stimulation.

Due to the use of vitrification technique and the appearance of the gonadotropins, physicians have been allowed to innovate the protocols applied to controlled ovarian hyperstimulation and have been able to obtain more oocytes in a shorter period for patients requiring rapid intervention, such as oncologic patients. Because of the accumulated experience with these new approaches, some investigators have recently proposed a double stimulation (DuoStim) protocol. Evidence of the competence of oocytes obtained from the luteal phase have been recently defined and published. Also, it has not been related with an increased risk for congenital anomalies.

The DuoStim is a protocol consisting of two stimulations within the same menstrual cycle, one in the follicular phase starting in day 2 of the cycle and the other in the luteal phase starting 5 days after the first ovarian puncture. Trigger is always performed with GnRH agonist.

Additionally, patients demanding infertility treatments are increasingly older and the use of preimplantation genetic testing (PGT) allows for a finer embryo selection along with better reproductive outcomes. Currently, most of PGTs are carried out at the blastocysts stage, which improve the prognosis but, on the contrary, also oblige to frozen those embryos and perform a deferred transfer, lengthening the procedure.

Another innovative tool for a more accurate embryo selection which has been recently described is the MitoScore. The MitoScore is a mitochondrial biomarker index developed by Igenomix aiming to indicate the energetic status of the embryo. It intends to select those embryos with best implantation potential and, therefore, more likely to result in an ongoing pregnancy after an IVF treatment. It is calculated dividing the number of mitochondrial DNA copies by the amount of nuclear DNA. Although still controversial, it has been proved by some authors to increase success rates of implantation and ongoing pregnancies in IVF cycles and to diminish the number of multiple gestations.

Since PGT is being more frequently requested from patients as women pursue infertility treatments at an advanced age with a poorer prognosis, sometimes physicians are compelled to perform several stimulation cycles to obtain more eggs and, consequently, a greater number of biopsied embryos. Hence, the idea of carrying out this study arises as an attempt to optimize each menstrual cycle to the maximum.

It is believed that the DuoStim protocol could be an alternative for this group of patients, allowing to obtain a larger number of oocytes in a shorter period, thus, increasing the number of biopsied embryos and possibly decreasing the interval to achieve a successful pregnancy.

The investigators aim to evaluate the potential usefulness of the DuoStim protocol for patients desiring to obtain oocytes as soon as possible. Also, using PGT, the investigators will compare the rate of euploid embryos per cycle in patients undergoing DuoStim protocol versus patients undergoing two conventional controlled ovarian hyperstimulation in consecutive cycles. Patients will include women with advanced age and poor response.

This is a unicentric, prospective, randomized, non-blind, parallel-group controlled phase IV clinical study. The investigators hypothesize that the rate of euploid embryos per cycle is similar in the DuoStim group compared to the group undergoing two conventional controlled ovarian hyperstimulation in consecutive cycles.

Furthermore the investigators will evaluate if there are differences regarding the number of total oocytes obtained, the number of mature oocytes, the number of biopsied blastocysts and the MitoScore index of the available euploid embryos. These variables will be assessed and compared depending on whether the oocytes were obtained in the follicular phase or the luteal phase for the DuoStim group. Resulting data will be compared with those obtained from the conventional stimulation group. The period elapsed from the beginning of the ovarian stimulation until the embryo transfer will also be addressed.

Patients will call the clinic at the Cycle Programing Department to arrange a treatment. After a short period taking contraceptive pills, patients will be referred to a medical appointment. At the time of the first consultation the attending physician will randomize patients desiring to participate and meeting inclusion criteria, using a random allocation software commissioned by the department of informatics. There will be no blinding since this study is an open trial.

Participants have the right to withdraw from the study at any time and for any reason without any inconvenience for their future medical care. Withdrawal means that the subject does not want to receive any further treatment nor does the patient wish to continue participating in the study. Reasons for withdrawal from the study: patient desire, lack of collaboration, toxicity or adverse event affecting patient's safety, decision of the principal investigator whenever the interruption is in favor of the patient's interests, death, and violation or breach of the study protocol.

The trial will be terminated when all participants have completed an adequate follow-up period. It might also be interrupted before completion date due to security reasons, failure to meet expected recruitment deadlines or even if there are any risks concerning patient's safety or health. All participants discontinued from the trial will remain in the follow-up phase, except for those who withdraw their informed consent or die.

Entries made in the Clinical Research Data Capture Profile (CRD) must be in accordance with those contained in the source documents. Data will be exported from the institutional repository software platform which withholds patient´s medical records. Integrity and accuracy will be checked by at least one investigator assuring that both extracted information and all the required regulatory documents are appropriate. Study files and all source documents will be stored for the time needed.

Considering an euploid embryo rate per cycle of 20% for conventional stimulation and a difference between means of 10% (Conventional X DuoStim group), a sample size of 136 patients (68 per arm) was estimated to obtain a power of 80% with an alfa error of 5%. A loss rate of 5% was also considered to calculate the sample size.

Categorical variables will be assessed by the number of subjects as well as absolute and relative frequencies. Continuous variables will be assessed by the means, medians, standard deviations, 25th and 75th percentiles, minimum and maximum. For both categorical and continuous variables, a confidence interval of 95% will be considered. The exploratory analysis of data will allow to determine quality of the data and to detect any abnormality.

The means and proportions of the descriptive variables will be compared to verify if the randomization was correctly performed. Whenever the variables are normally distributed, it will be applied a parametric test such as chi-square test for categorical variables and a T-student test or ANOVA for continuous variables. If the distribution is not normal a non-parametric test such as a Mann-Whitney U or Wilcoxon test will be applied according to the characteristics of the variable.

If the investigators find statically significant differences for descriptive variables between the two groups, those variables will be included in a regression model to control their interference.

Additionally, linear or logistic regression models will be defined, depending on whether the outcome variable is quantitative or categorical, respectively. It will allow to adjust possible confounding factors that may potentially influence the results.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* 35-42 years of age;
* Patients from the IVI Madrid undergoing controlled ovarian hyperstimulation cycle including PGT analysis for infertility treatment;
* BMI 18-30 kg/m2;
* Suspicion of suboptimal or poor response:

AMH < 1.5 ng/mL; AFC < 8; FSH > 10; Poor response in a previous cycle (defined as < 6 oocytes).

Exclusion Criteria:

* Simultaneous participation in another clinical trial or in any other study that could result in a confounding factor.

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Rate of euploid embryos per cycle | up to 9 months
  Rate of chromosomally normal embryos per cycle in the DuoStim group compared to the group undergoing two controlled ovarian hyperstimulation in consecutives cycles.

SECONDARY OUTCOMES:
Number of oocytes obtained | up to 9 months
  Total number of oocytes obtained in both arms after ovarian puncture
Number of fertilized oocytes | up to 9 months
  Number of fertilized oocytes in both arms after FIV/ICSI procedure
Number of biopsied blastocysts | up to 9 months
  Number of biopsied blastocysts in both arms
MitoScore index of the euploid embryos | up to 9 months
  Analysis of the MitoScore index of the euploid embryos obtained in both arms
Implantation rate | up to 9 months
  Implantation rate of euploid embryos in both arms after single or double embryo transfer
Pregnancy rate | up to 9 months
  Pregnancy rate of euploid embryos in both arms after single or double embryo transfer
Abortion rate | up to 9 months
  Abortion rate presented by each arm after single or double embryo transfer
Time until embryo transfer | up to 9 months
  Period elapsed from the beginning of the ovarian stimulation until the embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cerrillo, M.D., Ph.D., Principal Investigator — IVI Madrid
Locations (1):
- IVI Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baerwald AR, Adams GP, Pierson RA. A new model for ovarian follicular development during the human menstrual cycle. Fertil Steril. 2003 Jul;80(1):116-22. doi: 10.1016/s0015-0282(03)00544-2. PMID 12849812
- [Background] Cakmak H, Katz A, Cedars MI, Rosen MP. Effective method for emergency fertility preservation: random-start controlled ovarian stimulation. Fertil Steril. 2013 Dec;100(6):1673-80. doi: 10.1016/j.fertnstert.2013.07.1992. Epub 2013 Aug 26. PMID 23987516
- [Background] Cakmak H, Rosen MP. Random-start ovarian stimulation in patients with cancer. Curr Opin Obstet Gynecol. 2015 Jun;27(3):215-21. doi: 10.1097/GCO.0000000000000180. PMID 25919235
- [Background] Sonmezer M, Turkcuoglu I, Coskun U, Oktay K. Random-start controlled ovarian hyperstimulation for emergency fertility preservation in letrozole cycles. Fertil Steril. 2011 May;95(6):2125.e9-11. doi: 10.1016/j.fertnstert.2011.01.030. Epub 2011 Feb 3. PMID 21292255
- [Background] von Wolff M, Thaler CJ, Frambach T, Zeeb C, Lawrenz B, Popovici RM, Strowitzki T. Ovarian stimulation to cryopreserve fertilized oocytes in cancer patients can be started in the luteal phase. Fertil Steril. 2009 Oct;92(4):1360-1365. doi: 10.1016/j.fertnstert.2008.08.011. Epub 2008 Oct 18. PMID 18930226
- [Background] Bedoschi GM, de Albuquerque FO, Ferriani RA, Navarro PA. Ovarian stimulation during the luteal phase for fertility preservation of cancer patients: case reports and review of the literature. J Assist Reprod Genet. 2010 Aug;27(8):491-4. doi: 10.1007/s10815-010-9429-0. Epub 2010 May 9. PMID 20455017
- [Background] Kuang Y, Chen Q, Hong Q, Lyu Q, Ai A, Fu Y, Shoham Z. Double stimulations during the follicular and luteal phases of poor responders in IVF/ICSI programmes (Shanghai protocol). Reprod Biomed Online. 2014 Dec;29(6):684-91. doi: 10.1016/j.rbmo.2014.08.009. Epub 2014 Sep 6. PMID 25444501
- [Background] Ubaldi FM, Capalbo A, Vaiarelli A, Cimadomo D, Colamaria S, Alviggi C, Trabucco E, Venturella R, Vajta G, Rienzi L. Follicular versus luteal phase ovarian stimulation during the same menstrual cycle (DuoStim) in a reduced ovarian reserve population results in a similar euploid blastocyst formation rate: new insight in ovarian reserve exploitation. Fertil Steril. 2016 Jun;105(6):1488-1495.e1. doi: 10.1016/j.fertnstert.2016.03.002. Epub 2016 Mar 25. PMID 27020168
- [Background] Bentov Y, Esfandiari N, Gokturk A, Burstein E, Fainaru O, Casper RF. An ongoing pregnancy from two waves of follicles developing during a long follicular phase of the same cycle. Fertil Steril. 2010 Jun;94(1):350.e8-11. doi: 10.1016/j.fertnstert.2009.12.033. PMID 20138269
- [Background] Kuang Y, Hong Q, Chen Q, Lyu Q, Ai A, Fu Y, Shoham Z. Luteal-phase ovarian stimulation is feasible for producing competent oocytes in women undergoing in vitro fertilization/intracytoplasmic sperm injection treatment, with optimal pregnancy outcomes in frozen-thawed embryo transfer cycles. Fertil Steril. 2014 Jan;101(1):105-11. doi: 10.1016/j.fertnstert.2013.09.007. Epub 2013 Oct 23. PMID 24161646
- [Background] Chen H, Wang Y, Lyu Q, Ai A, Fu Y, Tian H, Cai R, Hong Q, Chen Q, Shoham Z, Kuang Y. Comparison of live-birth defects after luteal-phase ovarian stimulation vs. conventional ovarian stimulation for in vitro fertilization and vitrified embryo transfer cycles. Fertil Steril. 2015 May;103(5):1194-1201.e2. doi: 10.1016/j.fertnstert.2015.02.020. Epub 2015 Mar 23. PMID 25813280
- [Background] Diez-Juan A, Rubio C, Marin C, Martinez S, Al-Asmar N, Riboldi M, Diaz-Gimeno P, Valbuena D, Simon C. Mitochondrial DNA content as a viability score in human euploid embryos: less is better. Fertil Steril. 2015 Sep;104(3):534-41.e1. doi: 10.1016/j.fertnstert.2015.05.022. Epub 2015 Jun 11. PMID 26051102